CLINICAL TRIAL: NCT02412488
Title: Reveal LINQ™ In-Office 2 (RIO2) International Study
Brief Title: Reveal LINQ™ In-Office 2 (RIO2) Study International
Acronym: RIO2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: RIO2 International
Record Dates: First submitted 2015-04-06; First posted 2015-04-09 (Estimated); Results first posted 2019-02-11 (Actual); Last update posted 2019-02-11 (Actual); Status verified 2018-09

CONDITIONS: Arrhythmia
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Out of CathLab setting (Experimental): Out of cathlab insertion
  Interventions: Other: Out of cathlab insertion

INTERVENTIONS:
Other: Out of cathlab insertion — Insertion of the Reveal LINQ device in the "out-of-cathlab" setting (out of the operating room, cardiac catheterization or electrophysiology laboratory).

SUMMARY:
The purpose of the RIO 2 International study is to provide clinical and economic evidence to support moving the LINQ™ insertion procedure outside these traditional locations within the hospital, referred to as "out-of-cathlab".

DETAILED DESCRIPTION:
The traditional location of the LINQ™ insertion procedure is the catheterization laboratory, electrophysiology laboratory, or operating room. The purpose of the RIO 2 International study is to provide clinical and economic evidence to support moving the LINQ™ insertion procedure outside these traditional locations within the hospital, referred to as "out-of-cathlab".

ELIGIBILITY:
Inclusion Criteria:

* Patient is indicated for continuous arrhythmia monitoring with a Reveal LINQ™ Insertable Cardiac Monitor (ICM)
* Patient is at least 18 years of age or older if required by local regulations
* Patient is willing to undergo ICM insertion procedure outside of the cathlab, operating room, or EP lab setting with only local anesthetic
* Patient is willing and able to provide consent and authorize the use and disclosure of health information
* Patient is willing and able to comply with the elements of the clinical investigation plan including the required follow-up

Exclusion Criteria:

* Patient has unusual thoracic anatomy or scarring at the insertion site which may adversely affect the success of the insertion procedure
* Patient has reduced immune function or is otherwise at high risk for infection per physician discretion
* Current therapy with immunosuppressive agents or chronic steroid use e.g. Prednisone greater than 20mg per day
* Patient requires hemodialysis
* Patient with active malignancy or history of chemotherapy or radiation treatment
* Patient has had a recent (within 30 days) or an active infection including but not limited to pneumonia, urinary tract, cellulitis, or bacteremia
* Patient has had major surgery (in the past 6 months) Patient has undergone a procedure which required central venous or intra-arterial access (e.g. AF/VT ablation, EP study, coronary angiography) within the last 3 months or is scheduled for such a procedure while enrolled in the study
* Prior history of surgical infection, prosthetic device infection, or endovascular infection, including endocarditis, in the past 12 months
* Patient has a central venous port, an atrio-venous fistula, or a prosthetic valve
* Patient requires conscious or moderate sedation to receive LINQ™
* Patient already has an inserted or implanted loop recorder
* Patient is implanted or indicated for implant with a pacemaker, ICD, CRT device
* Patient is enrolled in another study that could confound the results of this study, without documented pre-approval from a Medtronic study manager
* Patient's life expectancy is less than 6 months
* Patient is legally incapable of giving consent
* Patient is pregnant* *Note: Possible pregnancy will be assessed by the physician asking the patient; a pregnancy test is not required

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 191 (Actual)
Dates: Start 2015-02; Primary Completion 2016-09-22 (Actual); Study Completion 2016-10-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: RIO2 Clinical Study Specialist, Study Chair — Medtronic

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sanders P, Piorkowski C, Kragten JA, Goode GK, Raj SR, Dinh T, Sohail MR, Anand R, Moya-Mitjans A, Franco N, Stromberg K, Rogers JD. Safety of in-hospital insertable cardiac monitor procedures performed outside the traditional settings: results from the Reveal LINQ in-office 2 international study. BMC Cardiovasc Disord. 2019 May 31;19(1):132. doi: 10.1186/s12872-019-1106-3. PMID 31151383

RESULTS

PARTICIPANT FLOW:
Groups:
- Out of CathLab Setting: The insertion of the Reveal LINQ device will be performed in the "out-of-cathlab" setting.
  Insertion of the Reveal LINQ device in the out of cathlab setting: Insertion of the Reveal LINQ device in the "out-of-cathlab" setting (out of the operating room, cardiac catheterization or electrophysiology laboratory).
Period: Overall Study
Arm/Group | Out of CathLab Setting
Started | 192
Reveal LINQ Implanted | 191
Completed | 174
Not Completed | 18
Not completed — Lost to Follow-up | 10
Not completed — Withdrawal by Subject | 5
Not completed — Physician Decision | 1
Not completed — No Reveal LINQ Insertion Attempt | 1
Not completed — Reveal LINQ explant | 1

BASELINE CHARACTERISTICS:
Population: Participants with Reveal LINQ Insertion Attempt
Arm/Group | Out of CathLab Setting
Number analyzed (Participants) | 191
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.8 (26.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 87
  Male | 104
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Australia | 34
  Canada | 28
  Germany | 28
  Italy | 15
  Netherlands | 32
  Spain | 35
  Sweden | 1
  United Kingdom | 15
Body Mass Index (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] | 27.9 (4.8)
Cardiomyopathy [Count of Participants; unit: Participants] | 10
Congestive Heart Failure [Count of Participants; unit: Participants] | 2
Hypertension [Count of Participants; unit: Participants] | 87
Myocardial infarction [Count of Participants; unit: Participants] | 3
Unexplained syncope [Count of Participants; unit: Participants] | 83
Diabetes [Count of Participants; unit: Participants] | 26
Renal dysfunction [Count of Participants; unit: Participants] | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Untoward Events
Description: An untoward event is a composite endpoint defined as a LINQTM or LINQTM insertion procedure related complication OR an unsuccessful LINQTM insertion procedure, where a LINQTM or LINQTM insertion procedure related complication is defined as an adverse event related to the LINQTM or a LINQTM insertion procedure resulting in:
  * Death
  * Termination of significant device function
  * Invasive intervention (e.g. includes LINQTM revision/explant for reasons other than diagnosis of underlying condition, intravenous drug administration)
Time Frame: 3 months
Population: Subjects exiting prematurely (prior to 3-month visit) without an untoward event were excluded from the primary analysis. There were 15 subjects exited prior to the 3-month visit all due to premature exit without having an untoward event
Measure: Count of Participants; unit: Participants
Arm/Group | Out of CathLab Setting
Number analyzed (Participants) | 176
Participants | 0
Statistical Analysis 1: Comparison: Out of CathLab Setting; There was no formal statistical hypothesis test associated with the primary outcome measure. Rather the goal of the primary study objective was to estimate the rate of untoward events associated with Reveal LINQ insertions performed in the "out-of-cathlab" setting through 3-months within a desired level of precision; Test type: Other — The goal of the primary study objective was to estimate the rate of untoward events associated with Reveal LINQ insertions performed in the "out-of-cathlab" setting through 3-months within a desired level of precision. The target sample size of approximately 200 subjects undergoing Reveal LINQ insertion was selected to ensure that the upper 95% confidence interval would be within 3 percentage points of the point estimate of the untoward event rate assuming the underlying rate was 2%; Event Rate expressed as a percent = 0, 95% CI 2-sided [0 to 2.1] — The estimate is the observed rate of untoward events expressed as a percentage. The 95% confidence interval is also expressed as a percentage

ADVERSE EVENTS:
Time Frame: All adverse events that were Reveal LINQ related, Reveal LINQ procedure related including any infections potentially resulting from the LINQ device or procedure as well as all serious events regardless of their relationship to the LINQ device or procedure were collected.
Description: An independent clinical events committee comprised of independent physicians who were not sponsor employees or study investigators adjudicated each reported event for its relationship to the Reveal LINQ system or procedure. All adverse event summaries are based on the clinical events committee's classification.
Arm/Group | Out of CathLab Setting
All-Cause Mortality (participants affected / at risk) | 0/191
Serious Adverse Events (participants affected / at risk) | 3/191
Other Adverse Events (participants affected / at risk) | 7/191
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Out of CathLab Setting (N=191)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
cerebrovascular accident (Nervous system disorders) | 1 (1)
syncope (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Out of CathLab Setting (N=191)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Implant site pain (General disorders) | 1 (1)
Incision site haemorrhage (Injury, poisoning and procedural complications) | 2 (2)
cerebrovascular accident (Nervous system disorders) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
This was a single arm study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes